CLINICAL TRIAL: NCT04468815
Title: An Open-Label Study to Assess Relative Bioavailability, Food Effect, and Esomeprazole Drug-Drug Interaction of BMS-986278 Tablets Following a Single Dose Administration in Healthy Participants
Brief Title: A Study to Assess the Levels in Blood Plasma of BMS-986278 in Healthy Participants Following Administration of Tablets, With or Without Food, and in the Presence of an Antacid (Esomeprazole)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM027-054
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: BMS-986278 suspension, fasted (Experimental)
  Interventions: Drug: BMS-986278 suspension
- Treatment B: BMS-986278 tablet, fasted (Experimental)
  Interventions: Drug: BMS-986278 Tablet
- Treatment C: BMS-986278 tablet, fed (Experimental)
  Interventions: Drug: BMS-986278 Tablet
- Treatment D: BMS-986278 tablet + esomeprazole capsule, fasted (Experimental)
  Interventions: Drug: BMS-986278 Tablet; Drug: Esomeprazole

INTERVENTIONS:
Drug: BMS-986278 Tablet — Specified dose on specified days
  Arms: Treatment B: BMS-986278 tablet, fasted; Treatment C: BMS-986278 tablet, fed; Treatment D: BMS-986278 tablet + esomeprazole capsule, fasted
Drug: Esomeprazole — Specified dose on specified days
  Other Names: NEXIUM
  Arms: Treatment D: BMS-986278 tablet + esomeprazole capsule, fasted
Drug: BMS-986278 suspension — Specified dose on specified days
  Arms: Treatment A: BMS-986278 suspension, fasted

SUMMARY:
The purpose of this study is to assess levels in blood plasma of BMS-986278 and the food effect in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations in the opinion of the investigator
* Women and men must agree to follow specific methods of contraception

Exclusion Criteria:

* Women of childbearing potential (WOCBP) and Women who are pregnant or breastfeeding
* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study
* Exposure to any investigational drug or placebo within 4 weeks of first study treatment administration.
* History of any significant drug and/or food allergies (such as anaphylaxis or hepatotoxicity)

Other protocol-defined inclusion/exclusion criteria apply

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of BMS-986278 | Up to 5 days
Area under the concentration-time curve from time 0 (dosing) to the time of the last quantifiable concentration observed (AUC(0-T) of BMS-986278 | Up to 5 days
Area under the concentration-time curve from time 0 (dosing) extrapolated to infinity AUC (INF) of BMS-986278 from the respective test treatments | Up to 5 days

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 29 days
Incidence of Serious Adverse (SAE's) | Up to 57 days
Incidence of AEs leading to discontinuation | Up to 29 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 48 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 48 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 48 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 48 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters | Up to 48 days
Incidence of clinically significant changes in physical examination findings | Up to 48 days
Incidence of clinically significant changes in clinical laboratory results: Clinical chemistry tests | Up to 48 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 48 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 48 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON (LPRA) - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm